CLINICAL TRIAL: NCT06592963
Title: Unfolding Severe and Enduring Eating Disorders (U-SEED)
Acronym: U-SEED
Status: Recruiting | Type: Observational
Sponsor: Uppsala University Hospital (Other)
Collaborators: The Söderström König Foundation (Unknown); Forte (Industry)
Responsible Party: Principal Investigator, Martina Isaksson, licensed psychologist, PhD, clinical researcher, Uppsala University Hospital
Other Study IDs: U-SEED
Record Dates: First submitted 2024-08-23; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Personality Disorders
Keywords: Registers; Severe and Enduring Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Personality Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — Samples retained, with potential for extraction of DNA from at least one of the types of samples retained (e.g., frozen tissue, whole blood)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main aim of this study is to identify biological and psychological characteristics as risk factors in individuals with severe and enduring eating disorders (SEED).

Specifically, the investigators aim to:

1. in a cohort of well-diagnosed eating disorder patients from 2005 followed up in National health registers, explore risk factors at baseline (recorded 2005-2007) for development of later SEED (the registry based cohort).
2. replicate the findings in a new sample of 50 adults with ongoing SEED. Participants will be assessed diagnostically and physically, and asked to fill out questionnaires and leave blood samples (the ongoing SEED sample compared with the register based cohort).
3. in a sample of 50 adults with SEED, explore demographic, biological, clinical, and psychological factors and examine the relation between these factors and symptom severity and functional impairment (the ongoing SEED sample).
4. explore participants perspectives on their symptoms and received care (the ongoing SEED sample).

DETAILED DESCRIPTION:
BACKGROUND, AIMS AND HYPOTHESES

Clinical factors such as psychiatric comorbidity and personality disorders, psychological and personality characteristics related to dysfunctional emotion regulation and loneliness, and biological factors such as dysregulation of the immune system, may all play a role in the developement, maintenance, and relapse of eating disorders. However, research in this field is scarce.

This projects aims is to increase our knowledge about risk factors for a severe course in eating disorders.

Hypotheses are:

* Personality disorders, comorbid psychiatric disorders and a high symptom load (generally and specifically for eating disorder symptoms) will be related to the development of SEED in the register based cohort
* The relation between SEED and personality disorders, comorbid psychiatric disorders and a high symptom load in the register based cohort will be replicated in the ongoing SEED sample
* In the ongoing SEED sample, symptom severity and functional impairment will be related to

  * Personality traits
  * Emotion dysregulation, maladaptive overcontrol and maladaptive undercontrol
  * Increased inflammation
  * More pronounced loneliness
  * Cognitive inflexibility

Primary outcomes are

* for aim 1: SEED at follow-up.
* for aim 2: factors identified from the register based study (aim 1). Thus, primary outcomes for aim 2 will be added to the protocol after analyses for aim 1 has been conducted.
* for aim 3: symptom severity and functional impairment
* for aim 4: patient perspectives of their symptoms and received care

Secondary outcomes are

* for aim 1: functional impairment, psychiatric and somatic comorbidity
* for aim 3: personality traits, emotion dysregulation, maladaptive overcontrol and maladaptive undercontrol, increased inflammation, more pronounced loneliness, cognitive inflexibility

PROCEDURE

The register based cohort: This adult cohort was consecutively recruited at the Eating Disorder Unit at the Uppsala Department of Psychiatry between 2005 and 2007. Of all 297 patients who came to the unit 218 (73%) participated. They were diagnosed according to gold standard including PD diagnoses, and thoroughly characterized in respect to clinical characteristics. They will be followed in national registries held by Statistics Sweden and the National Board of Health and Welfare, and these registers include the Swedish National Inpatient Register (IPR), the Longitudinal integrated database for health insurance and labour market studies (LISA) and the Registry of household statistics and the Swedish Medical Birth Register. By using registers both medical and social outcome can be examined. Factors from baseline can be related to outcome.

Tho ongoing SEED sample: Adult participants with SE-ED will be recruited through the ordinary staff that sees the participants at the Eating Disorder Unit at the Uppsala Department of Psychiatry combined with flyers and posters at the ED unit, through patient organizations, through the Uppsala University homepage, and through media. Those who themselves identify as having at least seven years duration of their ED and shown no or little response to treatment (SE-ED) who are interested in the study, will be guided to a web link were screening questions are provided. Inclusion criteria are having more than seven years of ED duration, having at least one evidence-based treatment without remission or resulting in relapse. Those completing the screening will be contacted, informed verbally in writing about the study and those fulfilling inclusion criteria will be invited to participate and sign an informed consent form. The investigators plan to include 50 participants. All participants will be invited to undergo a systematic diagnostic evaluation. The systematic evaluation consists of a clinical anamnestic history and three structured diagnostic interviews; either the MINI for DSM 5 or the Structured Clinical Interview for DSM-5 Axis I Disorders- Clinical Version (SCID-I CV) and Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5-PD) assessing personality disorders. Participants also undergo the Eating Disorder Examination interview (EDE). Participants are also weighed and measured. All diagnostic assessments are conducted by psychologists physicians or trained students, who have received training in the procedure and who are co-rated. Participants will also be asked about collection of biomarkers through Uppsala psychiatric patient samples (UPP), which is an infrastructure for the collection of biological materials at the Department of psychiatry at Uppsala University Hospital. All participants will be invited to take blood samples and inflammatory markers will be analyzed in accordance with the informed consent for UPP. After the structured evaluation, they will be interviewed about their perspectives on their symptoms and received care using a semi-structured interview guide. All interviews will be audio taped and transcribed verbatim.

DATA ANALYSES

For aim 1: Stratified Cox regression models will be estimated with year 2005 as entry time. Hazard ratios (HR) and corresponding 95% confidence intervals (CIs) will be calculated. Cumulative indices will be calculated and illustrated with Kaplan-Meier curves.

For aim 2: Descriptive statistics and generalized linear models will be performed comparing three groups: non-SEED and SEED from the register based cohort and SEED from the ongoing sample according to psychiatric symptoms, severity, comorbidity, personality disorders.

For aim 3: For the primary outcomes, generalized linear models will be used to analyze if more pronounced symptom severity and lower level of functioning will be explained by personality traits, emotion dysregulation, maladaptive overcontrol and maladaptive undercontrol, increased inflammation, more pronounced loneliness, cognitive inflexibility. Participants will be asked about collection of biomarkers through Uppsala Psychiatric Patient samples (UPP) (ethics approval Dnr 2012/081), which is an infrastructure for the collection of biological materials at the Department of Psychiatry at Uppsala University Hospital. All participants will be invited to participate in UPP and inflammatory markers will be analyzed in accordance with the informed consent for UPP. Inflammatory markers will be analyzed using an electrochemilumine scence sandwich immunoassay, Meso Scale Discovery (K15049D and K15198D, Rockville, MD, USA) a multiplex platform. For protein hormones, such as plasma adiponectin and leptin, a solid phase sandwich enzyme linked immunosorbent assay (ELISA) (Mercodia AB, Uppsala, Sweden) will be used. For the secondary outcomes, descriptive statistics will be presented.

For aim 4: Participant perspectives will be analysed qualitatively with thematic analyses

ELIGIBILITY:
For aim 1 (register based cohort):

Incl. criteria:

Attended care for eating disorders at Uppsala University Hospital between 2005 and 2007 and accepted to be included in a local quality register.

Excl. criteria: None

For aim 2 (ongoing SEED sample and register based cohort)

Incl. criteria:

* For ongoing SEED sample: Minimum age of 18, impairing eating disorder symptoms for at least seven years, and having at least one evidence-based treatment without remission or resulting in relapse.
* For register based cohort, see above.

Excl. criteria:

* For ongoing SEED sample: Eating disorders symptoms in need of emergency care, high risk for suicide, and an inability to respond to the questionnaires due to lack of knowledge in Swedish.

For aim 3 and 4 (the ongoing SEED sample). See above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The register based cohort:
  This adult cohort was consecutively recruited at the Eating Disorder Unit at the Uppsala Department of Psychiatry between 2005 and 2007. Of all 297 patients who came to the unit 218 (73%) participated in the study. They were diagnosed according to gold standard including PD diagnoses, and thoroughly characterized in respect to clinical characteristics.
  The ongoing SEED sample:
  Study population are individuals that themselves experience that their eating disorder have affected them in a significant way during at least the last seven years, who report having gone through at least one evidence-based treatment attempt, and that are willing to participate in the study. This adult sample will be recruited from the Eating Disorder Unit at the Uppsala Department of Psychiatry, via advertisement, through patient organizations, and through media. We plan to include 50 patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Eating disorder diagnosis during follow-up in registers (primary outcome for aim 1) | Registry data is retrieved autumn 2024
  Eating disorder diagnosis (AN, BN, BED, EDNOS, OSFED, UFED), collected from the National registries held by the National Board of Health and Welfare, from 2005 to 2024.
Findings identified from aim 1 - the register based study (primary outcome for aim 2) | Registry data is retrieved autumn 2024. Interviews and examinations performed with the ongoing SEED-sample for six hours.
  Primary outcome for aim 2 will be added to the protocol when the register study/aim 1 has been analysed, as the findings from those analyses will decide the primary outcome for aim 2.
Eating disorder examination interview (EDE-I) (Primary outcome for aim 3) | One hour
  EDE-I is a semi-structured interview for assessing symptoms of and diagnosing eating disorders. The EDE-I assesses a variety of eating disorder behaviors, weight control behaviors, and behavioral and cognitive features of eating disorder psychopathology.
Eating disorder Examination Questionnaire (EDE-Q) (Primary outcome for aim 3) | 20 minutes
  EDE-Q is a 28-item self-report questionnaire, designed to assess the range, frequency and severity of behaviors associated with an eating disorder. It is categorized into four sub-scales: Restraint, Eating Concern, Shape Concern and Weight Concern, and an overall global score. The score is obtained by calculating the mean for the total score and the subscales respectively (min = 0, max =6), higher scores indicate more severe eating disorder symptoms.
Clinical Impairment Assessment questionnaire (CIA) (Primary outcome for aim 3) | 10 minutes
  The CIA is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features, Each item is rated on a four-point Likert scale ranging from 'Not at all' to 'A lot'. The minimun score is zero and the maximum score is 48, with higher scores indicating a more severe impairment.
WHO Disability Assessment Schedule (WHODAS 2.0) (Primary outcome for aim 3) | 15 minutes
  WHODAS 2.0 measure individual dysfunction in six domains of daily activities (cognition, mobility, self-care, relationships with people, life activities, and participation). It is measured on a five-point Likert scale ranging from no difficulty, to extreme difficulty. The score is calculated by dividing the total score with the number of items, resulting in a minimum score of zero and maximum score of 4. Higher scores indicate higher disability.
Participants expressed views and experiences of their symptoms and received care (primary outcome for aim 4) | One hour
  A qualitative interview performed individually with each participant following a semi-structured interview guide.

SECONDARY OUTCOMES:
Functional impairment during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Demographic data describing level of education.
Functional impairment during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Demographic data describing civil status.
Functional impairment during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Demographic data describing number of children.
Functional impairment during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Demographic data describing occupation.
Functional impairment during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Demographic data describing level of income.
Functional impairment during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Demographic data describing welfare benefit.
Functional impairment during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Demographic data describing number of days in hospital care.
Functional impairment during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Demographic data describing compulsory care.
Psychiatric and somatic comorbidity during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Data describing psychiatric and somatic diagnosis.
Psychiatric and somatic comorbidity during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Data describing dental care.
Psychiatric and somatic comorbidity during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Data describing premature death.
Psychiatric and somatic comorbidity during follow-up in registers (secondary outcome for aim 1) | Registry data is retrieved autumn 2024
  Data describing cause of death.
The Mini-International Neuropsychiatric Interview (M.I.N.I) (secondary outcome for aim 3) | One hour
  M.I.N.I. is a structured diagnostic psychiatric interview designed to assess psychiatric disorders according to the DSM. It consists of a series of standardized questions and probes to elicit information about symptoms, duration, and severity of various psychiatric conditions such as mood disorders, anxiety disorders, substance use disorders, and psychotic disorders.
The Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5-PD) (secondary outcome for aim 3) | One hour
  Number, type and proportion of personality disorder diagnoses will be assessed by SCID-5-PD. It is a semistructured diagnostic interview for clinicians and researchers to assess the 10 DSM-5 Personality Disorders across Clusters A, B, C and Other Specified Personality Disorder. The SCID-5-PD includes the interview and the self-report screening questionnaire, the Structured Clinical Interview for DSM-5 Screening Personality Questionnaire (SCID-5-SPQ). SCID-5-SPQ will be used to screen for PDs before conducting the interview.
Blood pressure (secondary outcome for aim 3) | 30 minutes
  Blood pressure will be assessed with a valid and reliable device in a standardized procedure.
BMI (secondary outcome for aim 3) | 30 minutes
  Weight and height will be combined to report BMI in kg/m^2, assessed with a valid and reliable device in a standardized procedure.
EQ-Visual Analogue Scale (EQ-VAS) (secondary outcome for aim 3) | 5 minutes
  The EQ-VAS is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
The Avoidance and Fusion Questionnaire for Youth (AFQ-Y) (secondary outcome for aim 3) | 10 minutes
  The AFQ-Y is a self-rating instrument that measures psychological inflexibility. Participants rate their level of agreement on eight items on a 5-point Likert measuring one single factor. Score range is 0-24 and higher scores indicate a higher level of psychological inflexibility.
Social safeness and pleasure scale (SSPS) (secondary outcome for aim 3) | 10 minutes
  The SSPS is an 11-item self-rating instrument that assesses the extent to which people experience their world as safe, warm, and soothing, and how connected they feel to others. Participants indicate their answers on a five-point Likert scale, ranging from 1 (almost never) to 5 (almost all the time). Scores are added together to produce a total score in the range 11-55, with higher scores representing higher perceived social safeness and connectedness to others.
Loneliness scale (secondary outcome for aim 3) | 10 minutes
  The Loneliness scale is an 11-item self-rating instrument includes a 6-item emotional subscale and a 5-item social subscale. Respondents are presented with a series of statements and asked to indicate the extent to which the statement applies to their situation on a four-point Likert scale. The total score can range between 0-11 with higher scores indicating greater feelings of loneliness.
Demographic characteristics (secondary outcome for aim 3) | 10 minutes
  Gender, age, age at ED onset and treatment, and socio-demographic characteristics will be assessed.
Emotion Regulation Questionnaire (ERQ) (secondary outcome for aim 3) | 10 minutes
  The ERQ is a self-rating instrument designed to assess individual differences in the use of emotion regulation strategies. It is composed of ten items divided into two factors: cognitive reappraisal and expressive suppression. Participants indicate their answers on a 7-point Likert-scale ranging from 1 (total disagreement) to 7 (total agreement).
Ego Undercontrol Scale-13 (EUC-13) (secondary outcome for aim 3) | 10 minutes
  EUC-13 is a 13 item self-rating instrument designed to assess personality types based on how people inhibit or express their emotional impulses, identifying over- and undercontrolled personality styles. It is answered on a four-point Likert-scale ranging from Disagree very strongly to Agree very strongly. The total score can range between 1-4, with higher scores indicating higher undercontrol and lower scores indicating higher overcontrol.
Montgomery Åsberg Depression Scale (MADRS-S) (secondary outcome for aim 3) | 10 minutes
  MADRS-S is a 9-item widely used self-rating measure of depressive severity. The intention of the scale is to give an image of the patients current state of mind. The patient grades how he/she felt during the last three days. Items are rated on a seven-point Likert scale, providing a total score between 0-54, with higher scores reflecting greater depression severity.
UCLA Loneliness Scale (secondary outcome for aim 3) | 5 minutes
  UCLA Loneliness scale is a self-rating scale designed to measure ones subjective feelings of loneliness as well as feelings of social isolation. The scale comprises three questions that measure three dimensions of loneliness: relational connectedness, social connectedness and self-perceived isolation. Participants indicate their answers on a four-point Likert scale, providing a total score between 4-16, with higher scores indicating greater feelings of loneliness.
Swedish universities Scale of Personality (SSP) (secondary outcome for aim 3) | 20 minutes
  SSP is a self-report instrument assessing personality traits corresponding to biological correlates. It contains 91 items divided into 13 subscales. The scale can also be divided into a three-factor solution with Factor 1 reflecting Neuroticism; Factor 2 reflecting Aggressiveness; and Factor 3 reflecting Extraversion. Each item is given as a statement with a four-point response format, ranging from does not apply at all to applies completely. It is presented in standardized t-score ranging from 0-100 (mean 50 and standard deviation 10). Higher scorer indicate more pronounced characteristics of that specific trait.
Ghrelin (secondary outcome for aim 3) | 15 minutes
  Ghrelin will be analysed from blood samples. A solid phase sandwich enzyme linked immunosorbent assay (ELISA) (Mercodia AB, Uppsala, Sweden) will be used for the analyses.
Leptin (secondary outcome for aim 3) | 15 minutes
  Leptin will be analysed from blood samples. A solid phase sandwich enzyme linked immunosorbent assay (ELISA) (Mercodia AB, Uppsala, Sweden) will be used for the analyses
Adinopectin (secondary outcome for aim 3) | 15 minutes
  Adinopectin will be analysed from blood samples. A solid phase sandwich enzyme linked immunosorbent assay (ELISA) (Mercodia AB, Uppsala, Sweden) will be used for the analyses
Inflammatory markers (secondary outcome for aim 3) | 15 minutes
  Inflammatory markers will be analysed from blood samples. A panel of 100 different markers, will be anlyzed using an electrochemilumine-scence sandwich immunoassay, Meso Scale Discovery (K15049D and K15198D, Rockville, MD, USA) a multiplex platform.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University Hospital, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will not be made publicly available due to confidentiality but can be provided upon reasonable request.